CLINICAL TRIAL: NCT05050305
Title: A Phase 2 Study With Safety Run-In of Marizomib, Pomalidomide, and Dexamethasone For Relapsed and Refractory Multiple Myeloma and CNS Myeloma
Brief Title: Marizomib Central Nervous System (CNS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study support withdrawn
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Clifton Mo, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-551
Record Dates: First submitted 2021-04-14; First posted 2021-09-20 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma, Refractory; CNS Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — marizomib; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Marizomib plus pomalidomide and dexamethasone (Experimental): A safety run-in using a modified 3+3 dose de-escalation design with relapsed/refractory multiple myeloma (RRMM) cohort, expanded to a total of 16 participants once recommended phase 2 does (RP2D) has been identified.
  * Marizomib (MRZ) at a pre-determined dose on Days 1, 8, 15, 22 of a 28 day study cycle
  * Pomalidomide (POM) at a daily predetermined dose on Days 1-21 of a 28 day study cycle
  * Dexamethasone (DEX) at a daily predetermined dose on Days 1, 2, 8, 9, 15, 16, 22, 23 of a 28 day study cycle
  Simultaneously, relapsed/refractory multiple myeloma (RRMM) with central nervous system (CNS) involvement cohort will receive an identical modified 3+3 dose de-escalation design and expanded to an efficacy-evaluable total of 30 patients once recommended phase 2 does (RP2D has been identified
  Interventions: Drug: Marizomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Marizomib — Intravenous Infusion
  Other Names: Salinosporamide A
Drug: Pomalidomide — Taken orally
  Other Names: Pomalyst
Drug: Dexamethasone — Taken orally
  Other Names: Decadron; Dexasone; Hexadrol; Maxidex

SUMMARY:
This research is being done to test whether the investigational drug marizomib is safe and effective when used in combination with standard of care drugs for the treatment of multiple myeloma.

DETAILED DESCRIPTION:
This is a Phase 2 single-arm study, incorporating two cohorts and using the combination of marizomib plus pomalidomide and dexamethasone in relapsed/refractory multiple myeloma (RRMM) patients and in RRMM patients with CNS involvement.

This research study involves a three drug chemotherapy regimen which includes taking the study drug marizomib, as well as pomalidomide and dexamethasone. The U.S. Food and Drug Administration (FDA) has not approved marizomib as a treatment for any disease. The U.S. Food and Drug Administration (FDA) has approved pomalidomide and dexamethasone as a treatment option for multiple myeloma.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits. As the study is looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants that have multiple myeloma, not everyone who participates in this research study will receive the same dose of the study drug. The dose received will depend on the number of participants who have been previously enrolled in the study and how well participants have tolerated their doses. Participants will receive study treatment for as long as participants do not have serious side effects and their disease does not get worse.

It is expected that about 48 people will take part in this research study.

Bristol-Myers Squibb is supporting this research study by providing funding and study drug.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with MM based on standard IMWG criteria and currently requires treatment.
* Patients in the CNS-involved cohort must have CNS involvement of MM as defined by meningeal myelomatosis and/or radiological evidence of leptomeningeal disease and/or intracranial plasmacytoma involving brain parenchyma.
* Patients in the CNS-involved cohort must have received at least one or more previous lines of therapy including an IMiD and a proteasome inhibitor and have demonstrated disease progression on or within 60 days of completion of the last therapy.
* Patients in the RRMM cohort must have received at least two or more previous therapies including lenalidomide and a proteasome inhibitor and have demonstrated disease progression on or within 60 days of completion of the last therapy.
* Patients in the RRMM cohort must have measurable disease defined as at least one of the following:

  * Serum M protein ≥ 0.5 g/dL (≥5 g/L)
  * Urine M protein ≥200 mg/24 hours
  * Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
* Screening Laboratory evaluations within the following parameters

  * Absolute neutrophil count (ANC) ≥ 1,000 cells/dL (1.0 x 109/L) (Growth factors cannot be used within 14 days before first drug administration)
  * Platelet count ≥ 75,000 cells/dL (75 x 109/L) (without transfusions required during the 14 days prior to initiation of therapy)
  * Hemoglobin ≥ 8.0 g/dl (RBC transfusions are permitted)
  * Total Bilirubin ≤ 1.5 X upper limit of normal (ULN) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  * AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN
  * Calculated creatinine clearance ≥ 45 mL/min
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* All study participants must be registered into the mandatory POMALYST REMS® program, and be willing and able to comply with the requirements of the POMALYST REMS® program.
* Females of reproductive potential must adhere to the scheduled testing as required in the POMALYST REMS® program.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
* Patients have given voluntary written informed consent before performance of any study-related procedures not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior exposure to marizomib. and primary refractoriness to pomalidomide or a pomalidomide combination. Prior pomalidomide exposure is permitted but patients must have shown tolerance (defined as no grade 3 or greater non-hematologic toxicity), as well as responsiveness to pomalidomide-based therapy (defined as MR or better).
* Diagnosed or treated for another malignancy within 3 years prior to enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy/watchful waiting.
* Known GI disease or GI procedure that could interfere with the oral absorption of pomalidomide including difficulty swallowing.
* Systemic treatment, within 14 days before the first dose of pomalidomide, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
* Peripheral neuropathy ≥ Grade 3, or Grade 2 with pain on clinical examination during the screening period.
* Any medical or psychiatric illness that in the investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participating in this study.
* Current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, Grade 3 thromboembolic event or myocardial infarction within the past 6 months.
* The following therapies within the stated time frames prior to initiation of therapy: previous cytotoxic therapies, including cytotoxic investigational agents, for MM within 3 weeks; IMiDs, PIs, corticosteroids, other approved therapeutics and monoclonal antibodies (Mabs) within 2 weeks; and investigational therapies within 4 weeks. Please note consideration of the interval for investigational agents from already approved classes of drug in MM (e.g. Cell-Mods, Mabs) can be considered on a case by case basis with the PI. Prior peripheral stem cell transplant within 12 weeks and the use of live vaccines within 30 days.
* Prior allogeneic stem cell transplantation with active graft-versus-host-disease (grade 2 or greater).
* Prior major surgical procedure or radiation therapy within 4 weeks of initiation of therapy (this does not include limited course of radiation used for management of bone pain within 7 days of initiation of therapy).
* Daily requirement for corticosteroids equivalent to > 10 mg/day prednisone, except for inhalation corticosteroids, for the RRMM cohort. For patients with CNS involvement who require a higher dose of corticosteroids for control of vasogenic edema (e.g. 16 mg/day dexamethasone), eligibility will be determined on a case-by-case basis after discussion with the PI.
* Any > Grade 1 adverse reaction unresolved from previous treatments according to the National Cancer Institute - Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTC AE v.5.0). The presence of alopecia any grade or peripheral neuropathy ≤ Grade 2 without pain is allowed.
* Concurrent symptomatic amyloidosis or plasma cell leukemia.
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes).
* Known active infection requiring parenteral or oral anti-infective treatment within 7 days of start of therapy.
* Known human immunodeficiency virus or active hepatitis C viral infection.
* Active hepatitis B viral infection (defined as HBsAg+).

  * Patients with prior hepatitis B vaccine are permitted (defined as HBsAg-, Anti-HBs+, Anti-HBc-).
  * Non-active hepatitis B (HBsAg-, Anti-HBs+, Anti-HBc+) may be enrolled at the discretion of the investigator after consideration of risk of reactivation.
* Pregnant or breast-feeding females.
* Participants who are receiving any other investigational agents.
* History of erythema multiforme or severe hypersensitivity to prior IMiD's®.
* Inability to tolerate thromboprophylaxis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known hypersensitivity to thalidomide or lenalidomide or other drugs included in this study.

The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide, pomalidomide or similar drugs.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) Safety Run-In | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, up to 5 years
  MTD is defined as the highest dose level where no patients (of the 6 treated) develop a dose limiting toxicity (DLT)
Dose Limiting Toxicity (DLT) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, up to 5 years
  Toxicity summaries will be stratified by dose level, grade, and treatment attribution
The number and proportion of adverse events, graded as defined by CTCAE version 5.0. | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, up to 5 years
  CTCAE version 5.0.
Overall response rate (ORR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, up to 5 years
  Assessed using the updated International Myeloma Working Group Response Criteria (IMWG) (Rajkumar 2011).

SECONDARY OUTCOMES:
Time to response (TTR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, up to 5 years
  Assessed using the updated International Myeloma Working Group Response Criteria (IMWG) (Rajkumar 2011).
Progression free survival (PFS) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first. up to 5 years
  Assessed using the updated International Myeloma Working Group Response Criteria
Duration of response (DOR) | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, up to 5 years
  Assessed using the updated International Myeloma Working Group Response Criteria (IMWG) (Rajkumar 2011).
Overall survival (OS) | From date of enrollment until date of death from any cause, up to 5 years
  Assessed using the updated International Myeloma Working Group Response Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Mo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu